CLINICAL TRIAL: NCT01253317
Title: Pharmacological Treatment of Rett Syndrome by Stimulation of Synaptic Maturation With IGF-1
Brief Title: Treatment of Rett Syndrome With rhIGF-1 (Mecasermin [rDNA]Injection)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: International Rett Syndrome Foundation (Other); Autism Speaks (Other)
Responsible Party: Principal Investigator, Mustafa Sahin, Professor in Neurology, Harvard Medical School, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-08-0403
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Results first posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Rett Syndrome
Keywords: Rett Syndrome; IGF-1; Increlex; Mecasermin; IGF1; MECP2; RTT
MeSH Terms: conditions — Rett Syndrome | interventions — mecasermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rhIGF-1 (Experimental): Subjects will receive escalating twice-daily doses of IGF-1 over 4 weeks (40 µg/kg, 80 µg/kg, 120 µg/kg) and then continue treatment at 120 µg/kg BID for 20 weeks should they choose to enroll in the OLE.
  Interventions: Drug: rhIGF-1

INTERVENTIONS:
Drug: rhIGF-1 — 1) Multiple ascending dose (MAD) period (4 weeks): Subjects will receive escalating twice-daily doses of IGF-1 over 4 weeks (40 µg/kg, 80 µg/kg, 120 µg/kg) and then continue treatment at 120 µg/kg BID for 20 weeks should they choose to enroll in the open-label extension period.
  Other Names: Mecasermin (brand name Increlex)

SUMMARY:
The investigators are recruiting children for a research study using a medication known as IGF-1 (mecasermin or INCRELEX) to see if it improves the health of children with Rett syndrome (RTT). To participate in the study your child must be female, between the ages of 2 to 12 and have a genetic diagnosis (MECP2 deletion or mutation) of Rett Syndrome. As you may know, there is no treatment for this illness. Currently, the standard management of Rett syndrome is supportive, which means attempting to prevent complications and treatment of symptoms.

This study involves testing an investigational drug, which means that even though IGF-1 is approved by the Food and Drug Administration (FDA) for use in children, it has not been used before to treat Rett syndrome specifically. Information from this research will help determine whether the drug should be approved by the FDA in the future for the treatment of Rett Syndrome.

There are five major goals to this study:

1. As one of the features of Rett Syndrome is unstable vital signs, the investigators are trying to determine if IGF-1 has any effect on normalizing your child's pulse, blood pressure and breathing pattern.
2. The safety of IGF-1 in children with Rett syndrome. The study personnel will ask you to complete a medication diary and side effect reporting form on a regular basis. They will assist you in completing this by telephone interviews. Your child will undergo 2 lumbar punctures performed at the bedside in the clinical research facility. In addition, laboratory tests will be performed throughout the study to evaluate the safety of IGF-1. These will be blood tests similar to those provided in routine clinical care. Your child will undergo regular non-invasive comprehensive physical examinations including neurological and eye examination, tonsil evaluation, electrocardiograms (ECG), measurement of height, weight and head circumference.
3. IGF-1 may improve your child's behavior, communication and speech. In order to measure this, the investigators will evaluate your child once during each month of treatment with neurodevelopmental assessments and a neurological exam. Investigators will also ask you about her behavior and day-to-day functioning through a structured parental interview and questionnaires.
4. We will examine your child's cortical function through use of electroencephalography (EEG) in conjunction with presentation of visual and auditory stimuli. EEG is a non-invasive way of recording the electrical activity of your child's brain.
5. Children with Rett Syndrome sometimes experience "flushing" in their cheeks or have exceptionally cold hands or feet and/or abnormal perspiration. The Qsensor® is a non-invasive device worn on a fabric bracelet that continually measures your child's perspiration level and body temperature. We would like to use the Qsensor® to determine whether or not IGF-1 improves these symptoms.

   .

DETAILED DESCRIPTION:
There are two treatment periods in the trial. The multiple ascending dose (MAD) period is an intensive 4-week pharmacokinetic study which will require 3 inpatient stays and 4 half-day outpatient visits. During in-patient sessions, an IV line will be placed for frequent blood samples. A lumbar puncture will be performed by a physician at the beginning and again at the end of the MAD. The primary goal of the MAD is to determine the safety of IGF-1 therapy for girls with RTT. As such, the investigators will ask that you monitor your child's blood sugar levels using a glucometer. At the end of the MAD, you will have the option of enrolling your daughter in an additional 20 weeks of open-label IGF-1 treatment.

ELIGIBILITY:
Inclusion Criteria:

* female
* with RTT (typical or variant) as defined using the internationally agreed 2010 RettSearch criteria.
* genetically defined mutation or deletion of the MECP2 gene.
* Girls will have the following prepubertal status: (1) Tanner stage 1 or 2 breast development; (2) Tanner stage 1 or 2 pubic hair development; (3) and younger than 12 years by bone age.
* Chronological age must be 2 years or older

Exclusion Criteria:

* prior therapeutic use of IGF-1, growth hormone, Lupron® or sex steroids
* allergy to the trial product
* co-morbid or chronic illness beyond that known to be associated with Rett Syndrome: diabetes mellitus, fatty acid oxidation disorder, chromosomal aneuploidy, syndromes associated with high risk of malignancy, current or previous exposure to spinal irradiation or history of malignancy.
* severe scoliosis (defined as a spinal curve of 70 degrees or more as measured on clinical and radiological examination)

Ages: 2 Years to 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2010-12; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Sahin, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: International Rett Syndrome Foundation website — http://www.rettsyndrome.org/
- See also: Autism Speaks website — http://www.autismspeaks.org/
- See also: PNAS publication of phase 1 IGF-1 trial in RTT — http://www.ncbi.nlm.nih.gov/pubmed/24623853

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-label IGF-1 Treatment: Twelve girls with MECP2 mutations participated in the 4-week multiple ascending dose (MAD) period of open-label treatment with IGF-1 (mecasermin). The MAD focused on obtaining PK data, determining cerebrospinal fluid (CSF) penetration, evaluating safety and tolerability, and estimating feasibility of automated cardiorespiratory measures as biomarkers. Mecasermin was escalated over a 4-week period, beginning with twice daily injections of 40 mcg/kg the first week, 80 mcg/kg the second week, and 120 mcg/kg during the third and fourth weeks. CSF samples were obtained prior to initiating treatment and after completing the fourth week.
  10 of these subjects went on to complete the open label extension (OLE). The OLE was designed to obtain additional information on safety, tolerability, and cardiorespiratory measures after 20-weeks of treatment, as well as preliminary data on neurologic and behavioral parameters. During the 20-week OLE subjects were evaluated every 5 weeks.
Period: Overall Study
Arm/Group | Open-label IGF-1 Treatment
Started | 12
Completed | 10
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: Twelve girls with MECP2 mutations participated in the 4-week MAD period; ten of them continued and completed the subsequent 20-week OLE. Nine subjects met full diagnostic criteria for RTT, all of whom continued in the OLE.
Arm/Group | Open-label IGF-1 Treatment
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Time Frame: biweekly during the MAD and every five weeks during the OLE
Population: Subjects that had the same adverse event more than once are counted only one time using the closest relationship to study medication.
Measure: Number; unit: Adverse events
Groups:
- 4-week Multiple Ascending Dose (MAD): Twelve girls with MECP2 mutations participated in the 4-week multiple ascending dose (MAD) period of open-label treatment with IGF-1 (mecasermin). The MAD focused on obtaining PK data, determining cerebrospinal fluid (CSF) penetration, and evaluating safety and tolerability of IGF-1.
- 20-week Open Label Extension (OLE): 10 subjects that previously participated in the MAD went on to complete the OLE and were monitoring for safety of prolonged treatment (20 weeks).
Arm/Group | 4-week Multiple Ascending Dose (MAD) | 20-week Open Label Extension (OLE)
Number analyzed (Participants) | 12 | 10
Adverse events
  Unrelated adverse events | 4 | 4
  Possibly related adverse events | 2 | 17
  Probably related adverse events | 2 | 9

2. Primary Outcome: Pharmacokinetic (PK) Profile - Areas Under the Curve (AUCt)
Time Frame: 60 minutes pre-dose and 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 8.0, and 12.0 hours post-dose on days 1, 8, 15 and 29.
Measure: Mean (Standard Error); unit: ng.h/mL
Arm/Group | Open-label IGF-1 Treatment
Number analyzed (Participants) | 12
ng.h/mL
  Day 1: 40 mcg/kg dose | 2050.0 (235.2)
  Day 29: 120 mcg/kg dose | 3348.9 (261.9)

3. Secondary Outcome: Change From Pre-MAD Apnea Index at Post-OLE
Description: Apnea indices were compared from pre-MAD (prior to initiating treatment) to post-OLE (after 20 weeks of IGF-1 therapy). A negative value indicates a reduction in apnea index; representing an improved outcome. Apnea Index is defined as the number of apneas (≥ 10 seconds in length) occuring within one hour. The Apnea Index is calculated by dividing the number of qualifying apneic events by the number of hours in which they occurred. An apnea index greater than or equal to 5 is considered clinically significant by the American Academy of Sleep Medicine (AASM).
Time Frame: pre-MAD (baseline) to post-OLE (after 20 weeks of IGF-1 treatment)
Population: Two subjects enrolled in the MAD did not continue participation in the OLE and one subject was excluded from the analysis because, upon further medical record review, she did not meet diagnostic criteria for Rett syndrome.
Measure: Mean (Standard Error); unit: apneas per hour
Groups:
- MAD and OLE Treatment Periods: Twelve girls with MECP2 mutations participated in the 4-week multiple ascending dose (MAD) period of open-label treatment with IGF-1 (mecasermin). The MAD focused on obtaining PK data, determining cerebrospinal fluid (CSF) penetration, and evaluating safety and tolerability of IGF-1. Ten subjects that previously participated in the MAD went on to complete the OLE and were monitoring for safety of prolonged treatment (20 weeks).
Arm/Group | MAD and OLE Treatment Periods
Number analyzed (Participants) | 9
apneas per hour | -7.12 (4.58)

4. Secondary Outcome: Change in Social Avoidance Subscale Scores on the ADAMS From Pre-OLE to Post-OLE
Description: The Anxiety Depression and Mood Scale (ADAMS) is completed by the parent/caregiver and consists of 29 items which are scored on a 4-point rating scale that combines frequency and severity ratings. The Social Avoidance subscale [0 = best; 20 = worst] of the ADAMS is reported as a secondary outcome measure. A negative value indicates a decrease in the Social Avoidance subscale; which represents an improved outcome.
Time Frame: Pre-OLE (visit 1) and post-OLE (after 20 weeks of IGF-1 therapy)
Population: The ADAMS was not completed during the MAD.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- 20-week Open Label Extension (OLE): 10 subjects that previously participated in the MAD went on to complete the OLE and were monitored for safety of prolonged treatment (20 weeks).
Arm/Group | 20-week Open Label Extension (OLE)
Number analyzed (Participants) | 10
units on a scale | -1.44 (0.84)

ADVERSE EVENTS:
Time Frame: During the MAD and OLE (approximately 1 year, 4 months)
Description: AEs were assessed by guidelines published by the National Institutes of Health, National Cancer Institute, Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 Published: May 28, 2009 (v4.03: June 14, 2010)
Arm/Group | Open-label IGF-1 Treatment
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label IGF-1 Treatment (N=12)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) — During the MAD period, one serious adverse event occurred (respiratory distress) and was determined to be unrelated to the study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label IGF-1 Treatment (N=12)
Polydipsia (Endocrine disorders) | 6 (6) — Increased thirst
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Increased tonsil size
Snoring (Respiratory, thoracic and mediastinal disorders) | 5 (5) — Snoring
Vomiting (Gastrointestinal disorders) | 2 (5) — Vomiting
Salivary hypersecretion (Gastrointestinal disorders) | 2 (2) — Increased drooling
Nonscarring hair loss (Skin and subcutaneous tissue disorders) | 2 (2) — Hair loss
Precocious puberty (Reproductive system and breast disorders) | 4 (4) — Signs of early pubertal development

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes